CLINICAL TRIAL: NCT02265523
Title: The Effects of Exercise and Cycle Ergometry in Post-Operative Total Knee Patients-A Randomized Controlled Trial
Brief Title: Exercise and Cycle Ergometry Post TKA - A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Paolo Sanzo, Dr. Paolo Sanzo, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOAMA - Sanzo2014
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis; Deep Venous Thrombosis
Keywords: Arthroplasties, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Post-op Exercise Group (No Intervention): The standard post-operative exercises are already currently recommended to patients. Briefly, they include deep breathing and coughing, ankle pumping, buttock contractions, and static quadriceps strengthening. These are performed on a daily basis , 2-3 times per day, 30 repetitions.
- Viscus Group (Experimental): The Viscus (intervention) group will complete the standard post-operative exercises and will also have access to a Viscus V1.5 cycle ergometer 24 hours per day in their recovery room to use at their leisure.
  Interventions: Other: Cycle ergometer

INTERVENTIONS:
Other: Cycle ergometer — The Viscus V1.5 is a kinetic flywheel cycle ergometer that will allow participants' pedal revolutions to be tracked as well as time of use.
  Arms: Viscus Group

SUMMARY:
The purpose of this investigation is to examine the effect of, and improve patient compliance and motivation following total knee arthroplasty; to determine the efficacy of two post-surgical exercise programs on knee pain, function, range of motion, strength, and swelling (girth); and to establish a panel of biomarkers that will allow: a) early identification of patients at risk (i.e. unable to complete post-operative treatment) and; b) predict the likelihood of a successful treatment outcome post-surgically.

DETAILED DESCRIPTION:
Participants will be recruited from the current waiting list at either Thunder Bay Regional Health Sciences Centre or Big Thunder Orthopedics. The physician will be discussing the study and eligibility requirements with the potential participants. The research assistant at Big Thunder will then obtain signed consent from the potential participant during the pre-operative appointment. If the potential participant would like to discuss the study with the research team as well as the doctor before giving consent, the research team will be contacted. Adequate enrolment is expected as the amount of TKA performed in previous years has been above 300.

Eligibility screening will be performed by the physician in the surgeon's office prior to the potential participant giving informed consent. The physician will make the decision of whether or not someone is eligible based on examination of their medical history. If the potential participant is ineligible based on this information, they will not be involved in the study.

During a consultation, the physician will familiarize the potential participant with the study, the consent form, and any other relevant study material. The physician will answer any questions the potential participant has about the study and ask if they would rather speak with a member of the research team. The potential participant will be given the opportunity to discuss the study with an investigator and the Research Ethics Board prior to signing the consent form. If the participant wishes to consent to the study they will speak with the research assistant from Big Thunder at the pre-operative appointment who will obtain their signed consent form. The participant will be given a copy of the signed consent form and information letter for their records. The original form will be temporarily stored in a locked cabinet at Big Thunder, and picked up weekly to be retained by Dr. Paolo Sanzo in his locked office.

The two study groups will be the standard post-operative exercise protocol or the exercise protocol combined with the use of the Viscus V1.5 kinetic flywheel ergometer. The standard post-operative exercises are already currently recommended to patients. Briefly, they include deep breathing and coughing, ankle pumping, buttock contractions, and static quadriceps strengthening. The use of the kinetic flywheel ergometer will allow for pedal revolutions to be tracked as well as time of use. Participants randomized into the Viscus group will have access to a Viscus V1.5 24 hours per day in their recovery room to use at their leisure. All participants will track their own exercise in the exercise log which will be used to observe compliance. The participant's intensity of exercise will be rated on a 5-point Likert scale by the treating physiotherapist/nurse using the Sports Injury Rehabilitation Adherence Scale (SIRAS). The intensity of exercise will be rated from minimum effort to maximum effort; the frequency of exercise and the participants ability to follow instructions and advice will be rated from never to always; and the receptivity to changes in program will be rated from very unreceptive to very receptive.

Prior to surgery, demographic information such as height, weight, age and gender, as well as medical history and surgical history of the knee will be recorded.

Pain and Functional Measurements:

The following measures will be taken pre-operatively (day before surgery or at the pre surgery clinic), day 2 post-operatively, upon discharge, and 12 weeks post-operatively:

Knee pain will be measured using the visual analog scale (VAS). The VAS has a test-retest reliability of .71-.99, and a minimal clinically important difference of ±28 mm.

Functional status will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC has an internal consistency of .96; test-retest reliability of .64-.93; and is sensitive to change over time.

Knee swelling will be measured via girth measures taken 15 cm superior to the superior pole of the patella; at the supra and infrapatellar regions; and 15 cm inferior to the inferior pole of patella.

Knee flexion and extension ROM will be measured using a goniometer.

Resisted isometric knee flexion and extension strength will be measured with the subject lying supine and the knee positioned in the resting position (25° of flexion). The mean of three trials will be recorded in pounds using a Lafayette Manual Muscle Tester model 01165.

Motivation will be measured using the Behavioural Regulation in Exercise Questionnaire (BREQ2) pre- and post-operatively. This questionnaire will be given to the participants by the physiotherapist who takes the measures for VAS, WOMAC, girth and strength. This questionnaire was created by David Markland and Vannessa Tobin in 2004.

Adverse events such as DVT, PE, and wound infection will be recorded.

Blood markers:

Blood will be collected by a nurse trained in phlebotomy pre-operatively, 2 days post-operatively, and upon discharge. From the whole blood sample, samples will be prepared for plasma (von Willebrand factor) and serum (all remaining biomarkers, listed in the section below) following manufacturer's instructions. Plasma and serum will be isolated from whole blood, aliquoted, and stored at -80 degrees celsius until analysis using the enzyme-linked immunosorbent assays (ELISA) kits. Plasma and serum assays will be performed in Dr. Lees' lab at NOSM.

Panel of Biomarkers:

The panel of biomarkers is designed to screen for the following 3 categories:

Inflammation-The inflammatory markers were selected based on their potential to identify early infection complications (procalcitonin, IL-6). Recent research has established that procalcitonin is a highly specific rapid diagnostic marker of infection but will not give false positive values following surgical joint replacement. In addition, IL-6 has been linked to the risk of thrombogenic events and complications with recovery (fever, increased pain and decreased ROM).

Nutrition- It is estimated that 50-82% of patients in hospitals are undernourished which is linked to sub-optimal immune competence. The nutritional status biomarkers were selected based on their ability to identify both protein (prealbumin/transthyretin) and vitamin D status. The scientific literature related to vitamin D and bone health in older adults is extensive. It has been established that protein malnutrition is associated with impaired immune function. More recently vitamin D deficiency has also been shown to result in impaired immune function. Impaired immune function can manifest as post-operative infection and/or unsatisfactory rehabilitation. In addition, patients deficient in protein and vitamin D are known to be at risk of increased disability following THA and TKA and increased infection.

Thrombogenesis Risk- Deep venous thrombosis (DVT) with or without pulmonary embolism (PE) is a potentially life threatening complication of TKA surgery. Plasma von Willebrand factor predicts thromboembolic events. In addition, P-selectin is emerging as a promising biomarker of VT and high circulating levels of P-selectin have been established to be valuable as a predictor of VTE in cancer patients. Warfarin and aspirin therapies do not effect either plasma von Willebrand factor or soluble P-selectin.

During the consent process and throughout the study, if the participant or potential participant has difficulty understanding the English language, efforts will be made to provide translations for him or her.

The physiotherapist will obtain range of motion, strength, and girth measures, and will administer the VAS, WOMAC and BREQ2. This will occur while the participant is at the hospital. The physiotherapist or nurse will rate the participant's intensity of exercise based on a review of the exercise log book. A nurse trained in phlebotomy will draw the blood sample at the hospital and the research assistant will transport it back to NOSM where it will be aliquoted and labeled with the participant code, and stored at -80 degrees celsius until analysis.

Compiled measurements and dates each measurement was taken will be recorded on a data abstraction form by the physiotherapist or nurse who is taking the measurements.

The research team (Principal Investigator, Co-Investigators and research assistant) has access to all data. The research assistant will code this data in order to ensure confidentiality is kept in the case of samples/data leaving the hospital setting. Any non coded data will be stored at the hospital in a secure filing cabinet in a locked office. Computer data will be kept on a secure server on a password protected computer.

A nurse trained in phlebotomy will collect the blood samples. The research assistant, who has obtained the Transportation of Dangerous Goods certificate, will transport the sample from the hospital to NOSM for storage and analysis. For whole blood samples, samples will be prepared for PT and aPTT following manufacturer's instructions. For the serum biomarkers, serum will be isolated from whole blood 1.5 hours post draw, aliquoted, and stored at -80 degrees celsius until analysis using ELISA kits. All samples will be labeled with the participant code number as well as a letter for each time point. For example, A for pre-surgery, B for 2 days after surgery, and C for upon doscharge. Samples will be kept until all analysis is completed, after which all labels will be removed and samples will be disposed of as biohazardous waste.

Dr. Lees and the research assistant will be performing data analysis using ELISA kits on the blood samples at NOSM. Dr. Lees will be performing the statistical analysis portion at NOSM. Dr. Sanzo will be completing data analysis on the clinical and functional measurements at TBRHSC/SJCG. Missing data will have to be handled according to the type of data that is missing. For example, if some days are missing from the Viscus usage, these can be filled in due to the fact that total usage will be collected. We will still have total distance that included the day that was not recorded. If a blood sample was not collected, it will depend on the type of analysis. For analyses that depend on change (pre- versus post-), we will exclude that participant. However, the remaining blood samples for that participant could still be used in certain analyses (e.g., comparing group mean data for final day Viscus versus control). In addition, we would still be able to include all the functional and motivation data. There will be no interim analysis.

The target sample size is 100 participants total, with 50 in each group. With this group size, a power analysis performed on ROM measures (highest variability with the smallest change) with 10% potential change +/- 15% gives a power of 0.928. To achieve a power of 0.8, the minimum group size is 35 participants.

Repeated measures will be performed for individual improvements on pre-operative and post-operative measures. For measures that are independent of individual improvements, ANOVA will be used. A Fisher's LSD post hoc will be used to complete the analyses.

Along with quantitative methods, in order to measure compliance, the participant's intensity of exercise will be rated on a 5-point Likert scale by the treating physiotherapist/nurse using the Sports Injury Rehabilitation Adherence Scale (SIRAS). The intensity of exercise will be rated from minimum effort to maximum effort; the frequency of exercise and the participants ability to follow instructions and advice will be rated from never to always; and the receptivity to changes in program will be rated from very unreceptive to very receptive. Compliance will be taken into account in order to identify participants that may require additional monitoring to improve rehabilitative success.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50-80 years awaiting unilateral total knee arthroplasties
2. Willing to provide informed consent
3. Willing to be randomized to either of the post-operative treatment pathways and willing to follow the study protocol

Exclusion Criteria:

1. Serious cardiac, renal, hepatic, neoplastic and psychiatric diseases
2. Diabetes
3. Abnormal thyroid and adrenal function.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Knee pain/functional status/swelling/ROM/strength | All will be measured pre-operatively (baseline measure), and at day 2 post-operatively, upon discharge (anywhere from day 5-14 post-operatively), and 12 weeks post-operatively to observe changes from the baseline measure.
  Knee pain will be measured using the visual analog scale (VAS), and functional status will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Knee swelling will be measured via girth measures taken 15 cm superior to the superior pole of the patella; at the supra and infrapatellar regions; and 15 cm inferior to the inferior pole of patella, and flexion and extension ROM will be measured in degrees using a goniometer. The mean of three trials of resisted isometric knee flexor and extensor strength will be measured in lbs of force using a Lafayette Manual Muscle Tester.
Blood markers of inflammation/nutritional status/thrombogenesis risk | All will be measured pre-operatively (baseline measure), at day 2 post-operatively, and upon discharge (anywhere from day 5-14 post-operatively) to observe changes from the baseline measure.
  Plasma and serum will be isolated from whole blood samples and various assays will be completed to detect markers indicative of inflammation, poor nutritional status, and increased risk of thromboembolic events.

SECONDARY OUTCOMES:
Participant motivation. | Questionnaire will be completed pre-operatively, at day 2 post-operatively, upon discharge (anywhere from 5-14 days post-operatively), and 12 weeks post-operatively.
  Motivation will be measured using the Behavioural Regulation in Exercise Questionnaire (BREQ2) pre- and post-operatively.
Patient compliance. | Questionnaire will be completed pre-operatively, at day 2 post-operatively, upon discharge (anywhere from 5-14 days post-operatively), and 12 weeks post-operatively.
  Patient exercise intensity and compliance will be measured using the Sports Injury Rehabilitation Adherence Scale (SIRAS). The intensity of exercise will be rated from minimum effort to maximum effort on a 5 point Likert scale; the frequency of exercise and the participants ability to follow instructions and advice will be rated from never to always; and the receptivity to changes in program will be rated from very unreceptive to very receptive on this scale.

OTHER OUTCOMES:
Adverse events. | Will be completed from pre-operative to 12 weeks post-operatively as they arise.
  Adverse events such as deep vein thrombosis, pulmonary embolism, and wound infection will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

REFERENCES:
- [Derived] Sanzo P, Niccoli S, Droll K, Puskas D, Cullinan C, Lees SJ. The effects of exercise and active assisted cycle ergometry in post-operative total knee arthroplasty patients - a randomized controlled trial. J Exp Orthop. 2021 Jun 22;8(1):41. doi: 10.1186/s40634-021-00363-w. PMID 34159469